CLINICAL TRIAL: NCT00511810
Title: Evaluation of Omega-3 Fatty Acids as a Treatment-adjunct in Adolescent Patients With Major Depressive Disorder Exhibiting Partial Response to SSRI Medications: An Open-label Neuroimaging Trial
Brief Title: Omega-3 Fatty Acids as Adjunct Treatment for Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: The Inflammation Research Foundation (Other)
Responsible Party: Principal Investigator, Robert McNamara, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: McNamara Omega3 MDD
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Major Depressive Disorder
Keywords: Sadness; Insomnia; Loss of appetite; Fatigue; Trouble thinking
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders; Anorexia; Fatigue | interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose Fish Oil (Experimental): Capsule omega-3 fatty acids 2.4g/day (4 capsules/day)
  Interventions: Drug: Low Dose Fish Oil
- High Dose Fish Oil (Experimental): Liquid omega-3 fatty acid 15 g/day (2 tablespoons/day)
  Interventions: Drug: High Dose Fish Oil

INTERVENTIONS:
Drug: Low Dose Fish Oil — Omega-3 Fatty Acids 2.4g/day in capsule form (4 capsules per day)
  Other Names: OmegaRx - Zone Laboratories
  Arms: Low Dose Fish Oil
Drug: High Dose Fish Oil — Liquid omega-3 fatty acid 15 g/day (2 tablespoons/day)
  Other Names: OmegaRx - Zone Laboratories
  Arms: High Dose Fish Oil

SUMMARY:
The primary objective of the study was to determine the effects of 10-week adjunctive supplementation with 2 doses of LCn-3 fatty acids (fish oil) on cortical functional activity and biochemistry in adolescents with MDD.

The primary prediction was that LCn-3 fatty acid supplementation would dose-dependently increase prefrontal cortical functional activation during sustained attention and increase regional biochemical indices of cortical metabolism and integrity concentrations in association with reductions in depressive symptoms.

DETAILED DESCRIPTION:
This study is a 10-week open-label EPA+DHA treatment trial in adolescent (aged 12-18 years) patients with major depressive disorder exhibiting partial response to SSRI medications. After a screening visit, patients were randomized (stratified by gender) to open-label fish oil supplements at a fixed dose of either 2.4 g/day or 15 g/day (2 tablespoons/day) for 10 weeks.

A physical examination, a complete blood count (CBC), and thyroid stimulating hormone (TSH) levels were determined at baseline and Week 10, and vital signs (pulse, blood pressure, weight, height, body mass index, temperature) were obtained at each visit. At each visit, safety and tolerability were assessed using a structured side effect interview, the Side Effects Form for Children and Adolescents.

At baseline and all weekly visits, depression symptom severity was determined with the Children's Depression Rating Scale-Revised (CDRS-R), a 17-item observer-rated questionnaire, and remission was defined as a CDRS-R score of ≥28. If a patient's depressive symptoms worsened over the course of the trial (defined as 30% worsening relative to baseline on two consecutive visits using CDRS-R scores), they were withdrawn from the study. In view of the potential risk for developing hypomanic symptoms following LCn-3 fatty acid supplementation, manic symptom severity was monitored over the course of the trial with the Young Mania Rating Scale (YMRS), an 11-item observer-rated questionnaire.

fMRI scans were performed at baseline and at 10 weeks.

ELIGIBILITY:
Inclusion Criterion:

* Between the ages of 12-18 years.
* Diagnosis of MDD and not exhibited symptom remission CDRS-R (> 28 but < 40) despite being administered a standard therapeutic dose of an SSRI continuously for a minimum of 6 weeks.
* Ability and willingness to provide assent and informed, written consent from at least one biological parent.
* Present with biological parent or legal guardian.
* Willingness to maintain current dietary habits.
* Permission from treating physician
* Able to perform fMRI/MRS.

Exclusion Criterion:

* Inability or unwillingness to provide consent.
* Antecedent or concurrent serious medical illness.
* Clinically unstable medical disease, including cardiovascular, hepatic insufficiency, severe renal impairment, gastrointestinal, pulmonary, metabolic, endocrine, obesity or other systemic disease.
* History of seizures, excluding febrile seizures in childhood.
* Patients requiring treatment with any drug which might obscure the action of the study treatment.
* Female patients who are either pregnant or lactating.
* Clinically significant laboratory abnormalities in the last year on CBC or TSH tests.
* Judged clinically to be at suicidal risk (defined as having active suicidal ideation, intent or plan, or a serious suicide attempt within the past 6 months, or a baseline CDRS-R suicide score of >3).
* Hospitalized within the last 3 months
* Greater than 1 year outside appropriate age/grade level
* Pacemaker
* Cerebral aneurysm clip
* Cochlear implant
* Metal fragments lodged within the eye or braces
* Claustrophobia
* Necessity of sedation (no sedation will be given).
* History of loss of consciousness > 10 minutes in duration
* Allergy to seafood.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert McNamara, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in August, 2007 at the University of Cincinnati, Medical Sciences Building.
Pre-assignment Details: A total of 24 patients were screened and 20 patients met inclusion criteria.
Groups:
- High Dose Fish Oil: Liquid omega-3 fatty acid 15 g/day (2 tablespoons/day)
  High Dose Fish Oil : Liquid omega-3 fatty acid 15 g/day (2 tablespoons/day)
- Low Dose Fish Oil: Capsule omega-3 fatty acids 2.4g/day (4 capsules/day)
  Low Dose Fish Oil : Omega-3 Fatty Acids 2.4g/day in capsule form (4 capsules per day)
Period: Overall Study
Arm/Group | High Dose Fish Oil | Low Dose Fish Oil
Started | 8 | 12
Completed | 7 | 7 (2 terminated for worsening symptoms;1 refused a scan;2 lost to follow up (could not be contacted))
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Refused second scn | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Fish Oil | Low Dose Fish Oil | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 12 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (3.2) | 16.7 (2.9) | 15.0 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 20
Depression Score [Mean (Standard Deviation); unit: CDRS-R Score] — Patients were required to have a baseline score of >28 and <40 on the Children Depression Rating Scale-Revised (CDRS-R) despite being administered a standard therapeutic dose of an SSRI for a minimum of 6 weeks.
  CDRS-R Score | 33.5 (3.1) | 31.9 (6.5) | 32.7 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Mood Symptoms Ratings
Description: Depression symptom severity was determined with the Children's Depression Rating Scale-Revised (CDRS-R), which is a brief rating scale based on a semi-structured interview with the child. It is a 17-item observer-rated questionnaire where the 17 symptom areas are rated on a 6- or 7-point scale. Total score ranges from a low (not depressed) of 17 to a maximum (very depressed) of 108. Remission was defined as a CDRS-R score of <28. (The total score is the sum of the ratings on each of the 17 items.)
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: CDRS-R score
Groups:
- Baseline CDRS-R: High Dose Fish Oil: CDRS-R scores were computed for High Fish Oil groups.
- Baseline CDRS-R: Low Dose Fish Oil: CDRS-R scores were computed for Low Fish Oil groups.
Arm/Group | Baseline CDRS-R: High Dose Fish Oil | Baseline CDRS-R: Low Dose Fish Oil
Number analyzed (Participants) | 8 | 12
CDRS-R score | 33.0 (1.5) | 33.1 (1.7)

ADVERSE EVENTS:
Arm/Group | High Dose Fish Oil | Low Dose Fish Oil
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/12
Other Adverse Events (participants affected / at risk) | 0/8 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Fish Oil (N=8) | Low Dose Fish Oil (N=12)
Worsening of depressive symptoms (Psychiatric disorders) | 0 (0) | 2 (2) — Two patients in teh Low Dose Groupt experienced worsening of depressive symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes